CLINICAL TRIAL: NCT03757104
Title: Home-based Interventions to Test and Start (HITS): a Cluster-randomized Controlled Trial to Reduce Mortality and Incidence Through HIV Treatment
Brief Title: Home-based Intervention to Test and Start
Acronym: HITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Africa Health Research Institute (Other)
Collaborators: Heidelberg University (Other); University College, London (Other); London School of Hygiene and Tropical Medicine (Other); University of Glasgow (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Frank, Professor, Africa Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: A0001-BFC398/16
Record Dates: First submitted 2018-10-31; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: HIV; HIV Testing; Linkage to Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- micro-incentives (Experimental): micro-incentives only (8 communities)
  Interventions: Behavioral: micro-incentive
- EPIC-HIV (Experimental): Empowered through informed choice for HIV [male sensitive HIV specific decision support app] (males only in 8 communities)
  Interventions: Behavioral: EPIC-HIV
- micro-incentive and EPIC-HIV (Experimental): micro-incentives as well as EPIC [male sensitive HIV specific decision support app] (8 communities)
  Interventions: Behavioral: micro-incentive and EPIC-HIV
- control (No Intervention): standard of care

INTERVENTIONS:
Behavioral: micro-incentive — Residents in these communities are eligible to receive a R50 food voucher conditional on undergoing a home-based HIV test. If diagnosed with HIV, residents are eligible to receive a second R50 food voucher when they link to care within 6 weeks of the HIV test
  Other Names: Food voucher
  Arms: micro-incentives
Behavioral: EPIC-HIV — Men in these communities are eligible to receive a tablet-based male-sensitive HIV decision support app (EPIC-HIV 1)to encourage them to test for HIV at home. If diagnosed with HIV and do not link to care within a month of HIV test, they become eligible to receive a tablet-based male HIV specific decision support app (EPIC-HIV 2) to encourage them to link to HIV care.
  Arms: EPIC-HIV
Behavioral: micro-incentive and EPIC-HIV — micro-incentives: Residents in these communities are eligible to receive a R50 food voucher conditional on undergoing a home-based HIV test. If diagnosed with HIV, residents are eligible to receive a second R50 food voucher when they link to care within 6 weeks of the HIV test.
  EPIC-HIV 1:
  Men in these communities are eligible to receive a tablet-based male-sensitive HIV specific decision support app (EPIC-HIV 1) to encourage them to test for HIV at home. If diagnosed with HIV and do not link to care within a month of HIV test, they become eligible to receive a tablet-based male HIV specific decision support app (EPIC-HIV 2) to encourage them to link to HIV care.
  Other Names: Food Voucher and EPIC-HIV
  Arms: micro-incentive and EPIC-HIV

SUMMARY:
This study aims to establish the causal impact of two interventions - micro-incentives and a male-sensitive HIV- specific decision support app - on population-level HIV viral load and HIV-related mortality in men, as well as on population-based HIV incidence in young women.

DETAILED DESCRIPTION:
Research aim:

The primary aim of the home-based intervention to test and start (HITS) trial is to establish whether (i) the provision of two micro-incentives and (ii) a male-sensitive and HIV-specific decision support app will reduce population-level HIV viral load and HIV-related mortality in men, as well as population-level HIV incidence in young women.

Specific objectives

1. Establish the causal impact of two micro-incentives (aimed at increasing uptake of home-based HIV testing and linkage to care, respectively) on:

   1. Population-level HIV viral load in men
   2. Population-level HIV-related mortality in men
   3. Population-level HIV incidence in young women.
2. Establish the causal impact of a male-sensitive and HIV-specific decision- support app (called EPIC-HIV) on:

   1. Population-level HIV viral load in men
   2. Population-level HIV-related mortality in men
   3. Population-level HIV incidence in young women.
3. Establish the causal impact of the two conditional micro-incentives on:

   1. HIV status knowledge in men and women
   2. HIV knowledge in men and women
   3. HIV treatment knowledge in men and women
   4. HIV treatment utilization in men and women
   5. Sexual behavior in men and women
   6. Healthcare utilization in men and women
   7. Household healthcare expenditures
   8. Household wealth
   9. Retention in HIV care in men and women
4. Establish the causal impact of the male-sensitive HIV-specific decision support app on:

   1. HIV status knowledge in men and women
   2. HIV knowledge in men and women
   3. HIV treatment knowledge in men and women
   4. HIV treatment utilization in men and women
   5. Sexual behavior in men and women
   6. Healthcare utilization in men and women
   7. Household healthcare expenditures
   8. Household wealth
   9. Retention in HIV care in men and women

Hypothesis:

The investigators hypothesize that each of the two interventions - micro-incentives aimed at encouraging HIV testing and linkage to HIV care and a male-sensitive HIV-specific decision support app - will each increase HIV testing and HIV treatment uptake and via this mechanism lead to reduced population viral load and HIV-related mortality particularly in men. Reduced viral load among men, in turn, will reduce HIV incidence in young women.

Research design Following a formative phase to develop the design of the two HITS intervention the investigators will determine the causal impact of the interventions on our three primary endpoints in a 2x2 factorial cluster-randomized controlled trial with a baseline adjustment. A mixed- methods approach will be employed that combines the strengths of rapid formative social science research (that will inform the precise delivery of the HITS intervention) with a causally rigorous statistical methodology to evaluate the effectiveness of the HITS intervention.

The HITS intervention will be delivered through the Africa Health Research Institute's (AHRI) existing HIV surveillance operations. The investigators will randomize 45 communities to the four interventions. 8 communities each will receive one of the interventions (micro-incentives only, male-sensitive HIV-specific decision support app only); 8 communities will receive both interventions and 21 communities will receive standard-of-care. Communities will be stratified by incidence in young women (2004-2016) to derive a similar baseline incidence across intervention and standard-of-care communities prior to the implementation of the intervention. Both men and women will be eligible to receive the financial incentives to test and link to care, whilst only men will be eligible for the EPIC HIV-specific decision support application.

In the total of 3x8=24 communities in the intervention arms, an estimated total of 4,667 individuals will receive a HITS intervention. In the 21 communities, 4,900 individuals will receive the standard-of-care. Outcomes will be assessed in all eligible individuals living in the 45 communities, which together have an estimated population size of 30,000 adults.

Sample size calculation The study was powered using the outcome of HIV incidence in women aged 15-30. Using actual Africa Health Research Institute HIV incidence data, the investigators simulated the HITS intervention introduced in 2011 to 24 of the 45 communities in the study area. The investigators simulated an intervention that led to a 25% reduction in arm 1 (micro-incentives), 25% reduction in arm 2 (male-sensitive counselling) and a 32% reduction in the combined arm. Communities were stratified by baseline incidence (three strata) in young women (2004-2011) to allow for a similar baseline incidence in intervention and control communities and the investigators included a random effect in the simulations to adjust for clustering by community. The results show that the investigators would have been able to detect this reduction in incidence in >80% of simulation replicates (p<0.05). Therefore, if the investigators were to introduce the HITS intervention in 2018 and follow young women up for at least 3 years post intervention (ie utilize a total of 17 years of incidence data - 2004 to 2021) the investigators would be in excess of 90% powered to detect such a reduction in incidence in this critical age-group.

Research methodology Research site:

The trial will be managed from the Africa Health Research Institute, formerly Africa Centre that conducts a large longitudinal Demographic and Health surveillance. Participants will be enrolled during the routine HIV surveillance study (Population Intervention Program) - trained fieldworkers visit participants at home once a year to conduct household surveys using tablet computers and offer point of care HIV testing to all individuals aged 15+.

Study procedures:

In those arms of this cluster Randomized Controlled Trial (RCT) that include the once-off two-stage micro-incentive scheme, consenting men and women will be offered a first opportunity to earn a R50 food voucher (redeemable in a local supermarket) conditional on HIV testing. If a participant tests positive for HIV, he/she will have the opportunity to receive a second R50 food voucher conditional on linking within 6 weeks following the HIV test to one of the 11 local primary care clinics where HIV treatment and care are available.

In those arms of this cluster RCT that include the male-sensitive HIV-specific decision support app, men will be offered EPIC-HIV (a first version, so-called EPIC-HIV-1) prior HIV counseling and testing. EPIC-HIV-1 is aimed at increasing HIV testing uptake. Those participants who do not link to care within a month of the HIV test will be offered a second version of EPIC-HIV (so-called EPIC-HIV-2) at home to encourage linkage to care.

Follow up of participants:

Participants will be followed up routinely through the AHRI's ongoing population-based HIV surveillance. All participants will be followed up for at least 3 years.

Linkage to care will be routinely established via the AHRI's ongoing linkage of clinical records for all patients in the local public sector ART program in the demographic surveillance.

Data management: Data will be collected and managed by AHRI Research Data Management within PIP databases as per AHRI comprehensive study operating procedures (SOPs). The Population Intervention Platform (PIP) database has strictly restricted access via a data enclave on a secure server.

Data analysis:

All primary analyses (of both primary and secondary endpoints) will be intent-to-treat (ITT).

For the binary primary outcomes - HIV testing uptake, HIV treatment linkage, and population-level HIV viral suppression - the investigators will use generalized linear models with a Poisson distribution, log link function, and robust error terms to determine effect sizes (risk ratios).

For the two survival-analytical primary endpoints - population-level mortality among men and population-level HIV incidence among women - the investigators will use the Cox proportional hazards model to determine effect sizes (hazard ratios). If the proportional hazards assumption of the Cox model is violated, the investigators will use appropriate alternative survival analytical models.

In all primary analyses, the investigators will adjust for both baseline endpoints and clustering. For the survival analytical endpoints, the investigators will use data from the period 2004-2017 for baseline endpoint adjustment.

In addition, to the ITT analyses, the investigators will measure intervention effects adjusted for non-compliance using instrumental variable (IV) approaches

ELIGIBILITY:
Inclusion Criteria:

* 15 years old and above
* Resident members of households within the Population Intervention Platform
* Have consented to participate in Population Intervention Platform

additional eligibility criteria for EPIC-HIV

-Male

Exclusion Criteria:

* Refused to take part in Population Intervention Platform
* Participant reported to already be on ART

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4667 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV testing uptake at point of test offer in men | Baseline
  % received the rapid HIV test at home among those offered the test in men
HIV treatment linkage at 1 year in men | year 1
  % who visited study clinics and initiated antiretroviral therapy (ART) in men
Population-level HIV viral suppression in men | year 1
  Change in proportion with detectable viremia in men; HIV testing and viral load measurements are performed on the dried blood spot (DBS) samples collected during the annual survey
Population-level HIV-related mortality in men | year 3
  Change in HIV-related mortality rate measured as the number of HIV-related deaths per 1000 person-years of observation in men
Population-level HIV incidence in young women (15-30 years of age) | year 3
  Change in HIV incidence rate (number of HIV sero-conversions per 100 person-years of follow up) in young women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey

SECONDARY OUTCOMES:
HIV testing uptake at point of test offer in women | Baseline
  % received rapid HIV test at home among those offered the test in women
HIV treatment linkage at 1 year in women | year 1
  % who visited study clinics and initiated ART in women
Population-level HIV viral suppression (both sexes) | year 1
  Change in proportion with detectable viremia in both men and women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population-level HIV viral suppression (both sexes) | year 3
  Change in proportion with detectable viremia in both men and women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population-level HIV viral suppression in women | year 1
  Change in proportion with detectable viremia in women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population-level HIV viral suppression in women | year 3
  Change in proportion with detectable viremia in women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population-level HIV viral suppression in men | year 3
  Change in proportion with detectable viremia in men; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population level HIV incidence (both sexes) | year 3
  Change in HIV incidence rate (number of HIV sero-conversions per 100 person-years of follow up) in both men and women; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
Population-level HIV-related mortality (both sexes) | year 3
  Change in HIV-related mortality rate measured as the number of HIV-related deaths per 1000 person-years of observation in both men and women
Population-level all-cause mortality (both sexes) | year 3
  Change in all-cause mortality rate measured as the number of all-cause deaths per 1000 person-years of observation in both men and women
Population-level HIV-related mortality in women | year 3
  Change in HIV-related mortality rate measured as the number of HIV-related deaths per 1000 person-years of observation in women
Population-level HIV incidence in men | year 3
  Change in HIV incidence rate (number of HIV sero-conversions per 100 person-years of follow up) in men; HIV testing and viral load measurements are performed on the DBS samples collected during the annual survey
HIV status knowledge in men and women | year 1
  % ever received a test result for HIV in men and women
HIV prevention knowledge in men and women | year 1
  % reporting ever hearing about pre-exposure prophylaxis (PrEP)
HIV treatment utilization in men and women | year 1
  % reporting ever taking up ART for own health in men and women
Reported condom use in men and women | year 1
  % reporting condom use at last sex in men and women
Tuberculosis (TB) healthcare utilization in men and women | year 1
  % reported starting TB treatment in the past 12 months in men and women
Diabetes Healthcare utilization in men and women | year 1
  % reported starting diabetes treatment in the past 12 months
Hypertension healthcare utilization in men and women | year 1
  % reported starting blood pressure treatment in the past 12 months in men and women
Household wealth (household assets) | year 3
  Number of household assets (selected from a predefined list of 32 assets)
Household wealth (food security) | year 3
  % of adults in the household ever cutting the size of meals or missing meals due to insufficient money for food in the past 12 months
Partnership patterns in men and women | year 1
  % reporting having more than one sexual partner in the past 12 months in men and women
Retention in HIV care in men and women | year 1
  % who are retained in care (% patients having an ART clinic visit in previous 3 months) at 1 year post-initiation in men and women
Retention in HIV care in men and women | year 3
  % who are retained in care (% patients having an ART clinic visit in previous 3 months) at 3 years post-initiation in men and women
Patient viral suppression in men and women | year 1
  % who are remain virally suppressed (% patients where virus is undetectable) 1 year post-initiation in men and women
Patient viral suppression in men and women | year 3
  % who are remain virally suppressed (% patients where virus is undetectable) 3-years post-initiation in men and women

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tanser, PhD, Principal Investigator — Africa Health Research Institute
Locations (1):
- AHRI, Mtubatuba, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HY, Inghels M, Mathenjwa T, Shahmanesh M, Seeley J, Matthews P, Wyke S, McGrath N, Adeagbo O, Gareta D, Yapa HM, Zuma T, Dobra A, Blandford A, Barnighausen T, Tanser F. Effect of a Male-Targeted Digital Decision Support Application Aimed at Increasing Linkage to HIV Care Among Men: Findings from the HITS Cluster Randomized Clinical Trial in Rural South Africa. AIDS Behav. 2025 Jan;29(1):1-12. doi: 10.1007/s10461-024-04465-1. Epub 2024 Sep 11. PMID 39259239
- [Derived] Kim HY, Inghels M, Mathenjwa T, Shahmanesh M, Seeley J, Matthews P, McGrath N, Adeagbo O, Gareta D, Yapa HM, Zuma T, Dobra A, Barnighausen T, Tanser F. The impact of a conditional financial incentive on linkage to HIV care: Findings from the HITS cluster randomized clinical trial in rural South Africa. medRxiv [Preprint]. 2024 Mar 18:2024.03.15.24304278. doi: 10.1101/2024.03.15.24304278. PMID 38562873
- [Derived] Kim HY, Inghels M, Mathenjwa T, Shahmanesh M, Seeley J, Matthews P, Wyke S, McGrath N, Adeagbo O, Gareta D, Yapa HM, Zuma T, Dobra A, Blandford A, Barnighausen T, Tanser F. Effect of a male-targeted digital decision support application aimed at increasing linkage to HIV care among men: Findings from the HITS cluster randomized clinical trial in rural South Africa. medRxiv [Preprint]. 2024 Mar 18:2024.03.15.24304373. doi: 10.1101/2024.03.15.24304373. PMID 38562824
- [Derived] Makofane K, Kim HY, Tchetgen Tchetgen E, Bassett MT, Berkman L, Adeagbo O, McGrath N, Seeley J, Shahmanesh M, Yapa HM, Herbst K, Tanser F, Barnighausen T. Impact of family networks on uptake of health interventions: evidence from a community-randomized control trial aimed at increasing HIV testing in South Africa. J Int AIDS Soc. 2023 Aug;26(8):e26142. doi: 10.1002/jia2.26142. PMID 37598389
- [Derived] Tanser FC, Kim HY, Mathenjwa T, Shahmanesh M, Seeley J, Matthews P, Wyke S, McGrath N, Adeagbo O, Sartorius B, Yapa HM, Zuma T, Zeitlin A, Blandford A, Dobra A, Barnighausen T. Home-Based Intervention to Test and Start (HITS): a community-randomized controlled trial to increase HIV testing uptake among men in rural South Africa. J Int AIDS Soc. 2021 Feb;24(2):e25665. doi: 10.1002/jia2.25665. PMID 33586911